CLINICAL TRIAL: NCT04414189
Title: Clinical Validation of HostDx Sepsis™ on NanoString; a Prospective Observational Validation Trial
Status: Completed | Type: Observational
Sponsor: Inflammatix (Industry)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: INF-06
Record Dates: First submitted 2020-05-22; First posted 2020-06-04 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The blood sample collection materials for the HostDx Sepsis test (PAXgene Blood RNA tubes) will be collected. EDTA tubes for plasma measurements of procalcitonin and IL-6 will be collected. Collection tubes for serum samples to measure viral antibodies and/or viral titers (indicative of reactivation of viral infection) will also be collected. These will be stored locally and processed at a later time point dependent on needs, i.e. suspicion of viral reactivation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: Patients with suspected sepsis at the time of admission to the ICU
  Interventions: Diagnostic Test: HostDx Sepsis
- Arm B: Patients not currently suspected but at high risk for sepsis.
  Interventions: Diagnostic Test: HostDx Sepsis

INTERVENTIONS:
Diagnostic Test: HostDx Sepsis — Blood collection for mRNA analysis

SUMMARY:
This study will analyze HostDx Sepsis results from whole blood samples collected from patients with suspected sepsis or at risk for sepsis in the surgical ICU

ELIGIBILITY:
Inclusion Criteria:

Arm A

1. Age > 18 years
2. Suspected sepsis at the time of admission to the ICU
3. Direct admission from the ED to the ICU with suspected/proven sepsis.
4. Post-operative ICU admission after sepsis source control procedure
5. Inpatients admitted to the ICU from the ward with suspected sepsis onset.
6. Able to provide subject/proxy informed consent within 96h

Arm B

1. Age > 18 years
2. No suspicion of sepsis at the time of admission to the ICU but at high risk for subsequent sepsis onset
3. Non-trauma admission from the ED to the ICU
4. Post-operative ICU admission
5. Severe trauma admission from the ED (injury severity score >15, hemorrhagic shock, severe traumatic brain injury, and or severe chest trauma)
6. Inpatients admitted to the ICU from the ward for decompensation not initially suspected to be secondary to sepsis.
7. Able to provide subject/proxy informed consent within 96h

Exclusion Criteria:

1. Pre- or post-transplant patients
2. Patients admitted solely for airway monitoring, or vascular/flap check monitoring
3. Previous diagnosis of sepsis on index hospitalization.
4. Unable to provide informed consent within 96h
5. Previously enrolled in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects admitted to the surgical ICU with suspected sepsis or at high risk for subsequent sepsis onset.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-06-07 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Validate the diagnostic accuracy of HostDx Sepsis in a cohort of 360 hospitalized patients enrolled at time of suspicion of sepsis or at high risk for developing sepsis. | Time to enroll 360 subjects, process samples, and complete the follow-up, an average of 1 year
  Percentage of correctly identified patients with bacterial and/or viral infections using HostDx Sepsis compared to clinical adjudications using routine clinical, laboratory, and other findings
Validate the prognostic accuracy of HostDx Sepsis in a cohort of 360 hospitalized patients enrolled at time of suspicion of sepsis or at high risk for developing sepsis. | Time to enroll 360 subjects, process samples, and complete the follow-up, an average of 1 year
  Percentage of patients with correctly predicted outcomes using HostDx Sepsis (7-day organ support), and agreement between observed likelihood ratios and target likelihood ratios for the interpretation bands in HostDx Sepsis
Validate the prognostic accuracy of HostDx Sepsis in a cohort of 360 hospitalized patients enrolled at time of suspicion of sepsis or at high risk for developing sepsis. | Time to enroll 360 subjects, process samples, and complete the follow-up, an average of 1 year
  Percentage of patients with correctly predicted outcomes using HostDx Sepsis (CCI), and agreement between observed likelihood ratios and target likelihood ratios for the interpretation bands in HostDx Sepsis
Validate the prognostic accuracy of HostDx Sepsis in a cohort of 360 hospitalized patients enrolled at time of suspicion of sepsis or at high risk for developing sepsis. | Time to enroll 360 subjects, process samples, and complete the follow-up, an average of 1 year
  Percentage of patients with correctly predicted outcomes using HostDx Sepsis (30-day mortality), and agreement between observed likelihood ratios and target likelihood ratios for the interpretation bands in HostDx Sepsis
Validate the prognostic accuracy of HostDx Sepsis in a cohort of 360 hospitalized patients enrolled at time of suspicion of sepsis or at high risk for developing sepsis. | Time to enroll 360 subjects, process samples, and complete the follow-up, an average of 1 year
  Percentage of patients with correctly predicted outcomes using HostDx Sepsis (90-day mortality), and agreement between observed likelihood ratios and target likelihood ratios for the interpretation bands in HostDx Sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida College of Medicine, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No